CLINICAL TRIAL: NCT02837679
Title: Oncogeriatric Intervention and Follow-up at Home to Improve Quality of Life and the Possibility to Accomplish Cancer Treatment in Multimorbid Elderly
Brief Title: Oncogeriatric Intervention and Follow-up at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Marianne Ørum, MD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Onkogeriatri randomiseret
Record Dates: First submitted 2016-06-27; First posted 2016-07-19 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Neoplasms; Geriatric Assessment; Lung Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Geriatrics; Polypharmacy; Quality of Life
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Geriatric follow up
  Interventions: Other: Geriatric Follow up
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Geriatric Follow up
  Arms: Intervention

SUMMARY:
The study is a randomized study of patients living in four municipalities in Eastern Jutland. After geriatric assessment half of the patients will be offered a tailor-made intervention in their homes. The follow-up will last for at least 90 days and include treatment of the patients' multimorbidity, e.g. of dehydration, anaemia, infections, and malnutrition. The other half of the patients, the results of the assessment and recommendations will be given to the patients and their general practitioner.

The primary efficacy variables are accomplishment of planned cancer treatment, reduction of complications and admissions to hospital and increased quality of life,.

If geriatric assessment and a tailor-made follow-up result in a better quality of life with less complications and admissions the offer may be extended to a longer period, younger age groups and other cancer diagnoses.

DETAILED DESCRIPTION:
Cancer of the head and neck (HNC), lung (LC), upper gastrointestinal channel (CUGI) and colo-rectal cancer (CRC) accounts for approximately 40% of cancer incidence in elderly people (defined as ≥70 years) in Denmark (DK). The four cancers account for more than 50% of the annual cancer-related deaths in DK. Incidence and mortality of cancer increases with age. Comorbidity (simultaneous presence of several medical conditions) are more present in older cancer patients than in younger This means that older cancer patients are more vulnerable by physiological, psychological and social means than younger. Older cancer patients frequent develop side effects of cancer treatment than younger cancer patients.

Comprehensive Geriatric Assessment (CGA), is a comprehensive investigation and assessment of various aspects of a person's health, carried out by a multidisciplinary team in order to identify, quantify problems and follow up on the identified problems. CGA comprises collecting information on comorbidity, polypharmacy, physical, psychological and cognitive problems, nutritional status and social support. Problems in these areas implies a worse prognosis in terms of survival, response to treatment and side effects of cancer treatment .

CGA have shown to be able to identify novel health problems in about half of elderly patients with cancer. It has previously been shown that the focused palliative care of patients with lung cancer with a focus on optimization of medication and follow up on unresolved problems increases the quality of life, eases depressive symptoms and increases survival. CGA is shown to be an effective base for intervention in order to increase the survival of the elderly in general (with no known cancer), in order to increase the physical and cognitive status, and to reduce the need for changes in housing facilities. Geriatric intervention based on CGA called Comprehensive Geriatric Care (CGC).

Frailty is a condition that occurs as a result of declining physiological reserve, causing vulnerability to health stressors. One way of defining frailty is based on CGA, where patients are divided into "frail" "vulnerable/pre-frail" and "fit" by performing CGA :

Frail: patients who meet one or more of the following: dependence in Activities of Daily Living (ADL), severe comorbidity, cognitive dysfunction, depression, malnutrition, or more than 7 different fixed daily preparations on time for CGA, (multivitamin not included).

Fit patients: independent in ADL and Instrumental Activities of Daily Living (IADL), no or minimal comorbidity, Cognitively intact and no nutritional problems.

Vulnerable / pre-frail patients: Neither Fit nor frail. Frailty is a potentially reversible mode. It is known that elderly patients may develop frailty during cancer treatment.

From a previously conducted study of 217 elderly patients with HNC, LC, and CRC CUGI, we know that a large part of the patients are frail (52%) or vulnerable (35%). Only 13% are fit . But we do not know the effect of providing geriatric follow-up to this population with regards to complications of cancer treatment, including the ability to be able accomplish cancer treatment as planned and the possibility of reducing hospital stay.

A study carried out on patients discharged from the Emergency Department or Geriatric wards, have shown that it is possible to reduce the admission time by offering CGA related to admission and add follow-up with the CGC compared to only providing CGA for patients in the hospital. In the study, hospitalization was reduced by 55% It has not previously been shown if CGA in an outpatient setting and subsequent Geriatric follow up on the problems identified can reduce hospitalization time and increase the proportion who accomplish cancer treatment per protocol in older cancer patients until 1 status examination compared to patients who only get CGA in the outpatient setting, but do not get geriatric follow-up afterwards.

It's oncology practice at first outpatient attendance to define what type of cancer a patient must have, this includes both the type of treatment, the aim of treatment (neoadjuvant, adjuvant, curative or palliative (life-prolonging / palliative)), dose of treatment and duration of treatment before status examination.

Intervention CGC is an intervention that is tailored to the individual patient based on the problem areas identified by CGA and the problems that occur within 90 days of enrollment. It can include home visits, visits to Aarhus University Hospital (AUH) in outpatient settings, scheduled and on demand and telephone contact. Patients will be followed for 90 days of enrollment or until reference to specialized palliative care treatment or death. The geriatric intervention may consist of liquid treatment, blood transfusion, oral or intravenous antibiotic administration, oxygen therapy, pain management, social intervention, nutritional intervention and lifeline telephone number The geriatric intervention will be different from patient to patient. There may be many or few contacts of various kinds. During the 90 days the number and nature of contacts (telephone / attendance / home visits) will be recorded as the interventions that are performed will be registered (medication changes, social work, nutrition efforts and efforts to optimize Physical functioning) Contact between the oncogeriatric team and the patient can be taken at the initiative of oncogeriatric team, patient or relatives. The oncogeriatric team can initiate treatment or refer to another department, if necessary.

Controls For the control group, the result and the recommendations of the CGA, which has been given to patients regarding. for example medication changes, social intervention (eg. adaptation of home care), physical optimization for example. training and nutrition recommendations will be summarized for the patient and with the patient's acceptance sent to the practitioner. Otherwise, no follow-upis performed in the period by oncogeriatric team.

After 3 months, the intervention group and control Group are tested by CGA and quality of life questionnaires in order to compare with baseline results and comparing the control group with the intervention group.

Blinding It is not possible to blind subjects to randomization. Likewise, it is not possible to blind the geriatric team in charge of the follow-up for the result of the randomization. The person that test subjects after 3 months is blinded to the randomization. Oncologists do not get information about randomization.

ELIGIBILITY:
Inclusion Criteria:

70 years or older with cancer of the head and neck, upper gastro intestinal cancer, colo-rectal cancer or Lung cancer, refered to Aarhus University Hospital for evaluation regarding oncological treatment on the Oncology Department at Aarhus University

* Living in following municipalities: Odder (excl. of the island of Thunø), Faurskov, Skanderborg og Aarhus
* frail or vulnerable by CGA
* Signed informed consent. For incapacitated patients: informed consent by relatives

Exclusion Criteria:

* evaluated 'fit´ by CGA
* Referred to specialized palliative care at time of first visit at the Oncology department
* Do not wish to participate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of admittance to initial planned oncological treatment | An average of 12 weeks
  Oncological specialist evaluates if treatment is completed as planned or if eventual deviations are of minor or major character
Change in Quality of life (QoL) | 90 days
  Participants with a Mini-Mental State Examination (MMSE)-score of 25 and above are tested using European Organisation of Research and Treatment of Cancer (EORTC) Core Questionnaire (C30) in combination with Elderly questionnaire (ELD14).
Change in Quality of life | 90 days
  Participants with a Mini-Mental State Examination (MMSE)-score below 25 are tested using "Depression List"

SECONDARY OUTCOMES:
90-day survival | Within 90 days from first geriatric contact
  Are patients still alive 90 days after geriatric contact?
Physical performance, chair-stand-test | Changes in physical performance from first geriatric contact to 90 days after
  Physical performance is measured using chair-stand-test
Physical performance, Barthel-100 | Changes in physical performance from first geriatric contact to 90 days after
  Physical performance is measured using Barthel-100
Physical performance, FAQ-IADL | Changes in physical performance from first geriatric contact to 90 days after
  Physical performance is measured using Functional Activities Questionnaire (FAQ)-IADL
Length of hospital stay | Within 90 days from first geriatric contact
  Sum of hospital bed days in study period

OTHER OUTCOMES:
1-year mortality | Within 1 year from first geriatric contact
  time to death within 1 year from geriatric contact
3-year mortality | Within 3 year from first geriatric contact
  time to death within 3 years from geriatric contact
5-year mortality | Within 5 year from first geriatric contact
  time to death within 5 years from geriatric contact
Health costs per patient | Outcome measure will be assessed from time of first geriatric contact and 90 days on (0-90 days)
  Costs used per patient at the hospital, in home care, by the GP and the pharmacy within 90 days after Comprehensive Geriatric Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Ørum, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregersen M, Jensen K, Orum M. The impact of multidisciplinary geriatric follow-up on quality of life in older, non-surgical prefrail and frail patients with cancer A randomized controlled trial. J Geriatr Oncol. 2024 Nov;15(8):102069. doi: 10.1016/j.jgo.2024.102069. Epub 2024 Sep 16. PMID 39288507